CLINICAL TRIAL: NCT06746233
Title: Drug-Eluting Balloon or Drug-Eluting Stent in Acute Myocardial Infarction: A Randomized Controlled Trial
Acronym: BOOST-AMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Cardiovascular Diseases, Vojvodina (Other)
Responsible Party: Principal Investigator, Mila Kovacevic, Assistant Professor, MD, PhD, University of Novi Sad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICDVojvodina 1482-1/3
Record Dates: First submitted 2024-12-13; First posted 2024-12-24 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: ST Elevation Myocardial Infarction (STEMI)
Keywords: STEMI; DES; DCB
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drug coated balloon (DCB) (Experimental): Drug (paclitaxel) coated balloon (DCB) with concentration of 3 μg Paclitaxel per 1 mm2
  Interventions: Device: Drug (paclitaxel) coated balloon (DCB)
- Second generation of drug eluting stents (DES) (Active Comparator): Drug eluting stent (DES)
  Interventions: Device: Second-generation Drug Eluting Stent (DES)

INTERVENTIONS:
Device: Drug (paclitaxel) coated balloon (DCB) — In the experimental arm, a drug-coated balloon (DCB) with a concentration of 3 μg of Paclitaxel per 1 mm² will be used in patients with STEMI following successful lesion preparation (defined as residual stenosis ≤30%, TIMI flow grade 2-3, and absence of flow-limiting dissection). If the result after DCB treatment is unsatisfactory, a bailout drug-eluting stent (DES) will be implanted.
  Arms: Drug coated balloon (DCB)
Device: Second-generation Drug Eluting Stent (DES) — If the patient is randomized to the DES treatment arm, a second-generation drug-eluting stent (DES) will be implanted using standard techniques.
  Arms: Second generation of drug eluting stents (DES)

SUMMARY:
The objective of the study is to compare drug-coated balloon (DCB) with the gold standard drug-eluting stent (DES) in percutaneous coronary intervention (PCI) for patients presenting with ST-elevation myocardial infarction (STEMI).

Randomization will be performed after successful culprit-lesion preparation and confirmation that all angiographic entry criteria are met. Patients will be randomly assigned in a 1:1 fashion to receive either treatment with a Paclitaxel-coated balloon alone or second or third-generation DES.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years with a life expectancy of >1 year;
* Patients fulfilling criteria for STEMI (>20 min of chest-pain; At least 1 mm ST-elevation in at least two contiguous leads, a new left bundle branch block or a true posterior myocardial infarction confirmed by ECG or echocardiography; Reperfusion is expected to be feasible within 12 h after onset of symptoms)
* Infarct related artery eligible for primary PCI (De novo lesion in a native coronary artery; Reference-vessel diameter ≥2.5 mm and ≤ 4 mm; Absence of severe calcification; Residual diameter stenosis of ≤30% (by visual assessment) after lesion preparation after lesion preparation; Absence of coronary dissection type ≥C.

Exclusion Criteria:

* Killip class>II on admission
* Known contraindication for aspirin, clopidogrel, ticagrelor, heparin or GP IIb/IIIa inhibitor
* Previous myocardial infarction
* Previous PCI in the territory of the infarct-related artery (IRA)
* Previous CABG
* 3-vessel disease requiring revascularization
* Left-main disease
* Extremely angulated or severely calcified vessels
* History of ischemic stroke within the past 6 months or hemorrhagic stroke
* Planned CABG for a non-culprit vessel
* Participation in another investigational trial that has not completed its primary endpoint or could interfere with the endpoints of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 598 (Estimated)
Dates: Start 2024-12-25 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
DoCE (Device-oriented composite endpoint) | 1 year and 2 years
  DoCE: A composite endpoint consisting of cardiac mortality, non-fatal target vessel myocardial infarction (NF-TVMI), and target lesion revascularization (TLR).

SECONDARY OUTCOMES:
Individual components of the primary endpoint (DoCE) | 1 year and 2 years
  Individual components of the primary endpoint (DoCE):
  * Cardiac mortality
  * Non-fatal target vessel myocardial infarction (NF-TVMI)
  * Target lesion revascularization (TLR)
Patient-oriented composite endpoint (PoCE) | 1 year and 2 years
  PoCE: Defined as a composite of all-cause death, any stroke, any myocardial infarction (MI), and any clinically or physiologically indicated revascularization.
Target vessel revascularization (TVR) | 1 year and 2 years
Target vessel failure (TVF) | 1 year and 2 years
  Target Vessel Failure (TVF): Defined as a composite of cardiac death, target vessel myocardial infarction (MI), and clinically or physiologically indicated target vessel revascularization (TVR).
BARC (Bleeding Academic Research Consortium) type 3 and 5 bleeding complications. | 1 year and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mila Kovačević, MD, PhD, Principal Investigator — Institute of Cardiovascular Diseases of Vojvodina
Locations (4):
- Serbia (4):
  - University Clinical Centre of Nis, Niš, Serbia
  - University Clinical Center of Serbia, Belgrade
  - Institute of Cardiovascular Diseases of Vojvodina, Kamenitz
  - University Clinical Center of Kragujevac, Kragujevac

REFERENCES:
- [Background] Scheller B, Eccleshall S. Drug-coated balloons for acute coronary syndromes. EuroIntervention. 2024 Jul 1;20(13):e791-e792. doi: 10.4244/EIJ-E-24-00019. No abstract available. PMID 38949238
- [Background] Byrne RA, Rossello X, Coughlan JJ, Barbato E, Berry C, Chieffo A, Claeys MJ, Dan GA, Dweck MR, Galbraith M, Gilard M, Hinterbuchner L, Jankowska EA, Juni P, Kimura T, Kunadian V, Leosdottir M, Lorusso R, Pedretti RFE, Rigopoulos AG, Rubini Gimenez M, Thiele H, Vranckx P, Wassmann S, Wenger NK, Ibanez B; ESC Scientific Document Group. 2023 ESC Guidelines for the management of acute coronary syndromes. Eur Heart J Acute Cardiovasc Care. 2024 Feb 9;13(1):55-161. doi: 10.1093/ehjacc/zuad107. No abstract available. PMID 37740496
- [Background] Merinopoulos I, Gunawardena T, Corballis N, Bhalraam U, Reinhold J, Wickramarachchi U, Maart C, Gilbert T, Richardson P, Sulfi S, Sarev T, Sawh C, Wistow T, Ryding A, Mohamed MO, Perperoglou A, Mamas MA, Vassiliou VS, Eccleshall SC. Assessment of Paclitaxel Drug-Coated Balloon Only Angioplasty in STEMI. JACC Cardiovasc Interv. 2023 Apr 10;16(7):771-779. doi: 10.1016/j.jcin.2023.01.380. PMID 37045498
- [Background] Fang Z, Ji J, He S, Liu N, Xu B. Drug-Coated Balloon vs. Drug-Eluting Stent in Acute Myocardial Infarction: A Systematic Review and Updated Meta-Analysis. Anatol J Cardiol. 2023 Jul 1;27(8):444-452. doi: 10.14744/AnatolJCardiol.2023.2953. Epub 2023 Jun 15. PMID 37329115
- [Background] Wang Z, Yin Y, Li J, Qi W, Yu B, Xu Z, Zhu W, Yang F, Cao M, Zhang H. New Ultrasound-Controlled Paclitaxel Releasing Balloon vs. Asymmetric Drug-Eluting Stent in Primary ST-Segment Elevation Myocardial Infarction - A Prospective Randomized Trial. Circ J. 2022 Mar 25;86(4):642-650. doi: 10.1253/circj.CJ-21-0315. Epub 2021 Nov 10. PMID 34759131
- [Background] Hao X, Huang D, Wang Z, Zhang J, Liu H, Lu Y. Study on the safety and effectiveness of drug-coated balloons in patients with acute myocardial infarction. J Cardiothorac Surg. 2021 Jun 21;16(1):178. doi: 10.1186/s13019-021-01525-8. PMID 34154628
- [Background] Vos NS, Fagel ND, Amoroso G, Herrman JR, Patterson MS, Piers LH, van der Schaaf RJ, Slagboom T, Vink MA. Paclitaxel-Coated Balloon Angioplasty Versus Drug-Eluting Stent in Acute Myocardial Infarction: The REVELATION Randomized Trial. JACC Cardiovasc Interv. 2019 Sep 9;12(17):1691-1699. doi: 10.1016/j.jcin.2019.04.016. Epub 2019 May 21. PMID 31126887
- [Background] Gobic D, Tomulic V, Lulic D, Zidan D, Brusich S, Jakljevic T, Zaputovic L. Drug-Coated Balloon Versus Drug-Eluting Stent in Primary Percutaneous Coronary Intervention: A Feasibility Study. Am J Med Sci. 2017 Dec;354(6):553-560. doi: 10.1016/j.amjms.2017.07.005. Epub 2017 Jul 19. PMID 29208251
- [Background] Jeger RV, Farah A, Ohlow MA, Mangner N, Mobius-Winkler S, Leibundgut G, Weilenmann D, Wohrle J, Richter S, Schreiber M, Mahfoud F, Linke A, Stephan FP, Mueller C, Rickenbacher P, Coslovsky M, Gilgen N, Osswald S, Kaiser C, Scheller B; BASKET-SMALL 2 Investigators. Drug-coated balloons for small coronary artery disease (BASKET-SMALL 2): an open-label randomised non-inferiority trial. Lancet. 2018 Sep 8;392(10150):849-856. doi: 10.1016/S0140-6736(18)31719-7. Epub 2018 Aug 28. PMID 30170854
- [Background] Tang Y, Qiao S, Su X, Chen Y, Jin Z, Chen H, Xu B, Kong X, Pang W, Liu Y, Yu Z, Li X, Li H, Zhao Y, Wang Y, Li W, Tian J, Guan C, Xu B, Gao R; RESTORE SVD China Investigators. Drug-Coated Balloon Versus Drug-Eluting Stent for Small-Vessel Disease: The RESTORE SVD China Randomized Trial. JACC Cardiovasc Interv. 2018 Dec 10;11(23):2381-2392. doi: 10.1016/j.jcin.2018.09.009. PMID 30522667
- [Background] Indermuehle A, Bahl R, Lansky AJ, Froehlich GM, Knapp G, Timmis A, Meier P. Drug-eluting balloon angioplasty for in-stent restenosis: a systematic review and meta-analysis of randomised controlled trials. Heart. 2013 Mar;99(5):327-33. doi: 10.1136/heartjnl-2012-302945. Epub 2013 Jan 18. PMID 23335497
- [Background] Kawai T, Watanabe T, Yamada T, Morita T, Furukawa Y, Tamaki S, Kawasaki M, Kikuchi A, Seo M, Nakamura J, Tachibana K, Kida H, Sotomi Y, Sakata Y, Fukunami M. Coronary vasomotion after treatment with drug-coated balloons or drug-eluting stents: a prospective, open-label, single-centre randomised trial. EuroIntervention. 2022 Jun 3;18(2):e140-e148. doi: 10.4244/EIJ-D-21-00636. PMID 34757917
- [Background] Kleber FX, Schulz A, Waliszewski M, Hauschild T, Bohm M, Dietz U, Cremers B, Scheller B, Clever YP. Local paclitaxel induces late lumen enlargement in coronary arteries after balloon angioplasty. Clin Res Cardiol. 2015 Mar;104(3):217-25. doi: 10.1007/s00392-014-0775-2. Epub 2014 Oct 28. PMID 25349065
- [Background] Ann SH, Balbir Singh G, Lim KH, Koo BK, Shin ES. Anatomical and Physiological Changes after Paclitaxel-Coated Balloon for Atherosclerotic De Novo Coronary Lesions: Serial IVUS-VH and FFR Study. PLoS One. 2016 Jan 29;11(1):e0147057. doi: 10.1371/journal.pone.0147057. eCollection 2016. PMID 26824602
- [Background] Madhavan MV, Kirtane AJ, Redfors B, Genereux P, Ben-Yehuda O, Palmerini T, Benedetto U, Biondi-Zoccai G, Smits PC, von Birgelen C, Mehran R, McAndrew T, Serruys PW, Leon MB, Pocock SJ, Stone GW. Stent-Related Adverse Events >1 Year After Percutaneous Coronary Intervention. J Am Coll Cardiol. 2020 Feb 18;75(6):590-604. doi: 10.1016/j.jacc.2019.11.058. PMID 32057373
- [Background] De Luca G, Damen SA, Camaro C, Benit E, Verdoia M, Rasoul S, Liew HB, Polad J, Ahmad WA, Zambahari R, Postma S, Kedhi E, Suryapranata H; Collaborators. Final results of the randomised evaluation of short-term dual antiplatelet therapy in patients with acute coronary syndrome treated with a new-generation stent (REDUCE trial). EuroIntervention. 2019 Dec 6;15(11):e990-e998. doi: 10.4244/EIJ-D-19-00539. PMID 31422929
- [Background] Keeley EC, Boura JA, Grines CL. Primary angioplasty versus intravenous thrombolytic therapy for acute myocardial infarction: a quantitative review of 23 randomised trials. Lancet. 2003 Jan 4;361(9351):13-20. doi: 10.1016/S0140-6736(03)12113-7. PMID 12517460